CLINICAL TRIAL: NCT01545037
Title: Effect of Lactobacillus Acidophilus CL1285®, L. Casei LBC80R® and L. Rhamnosus CLR2® on Symptoms of Irritable Bowel Syndrome: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: Effect of BIO-K+ on Symptoms of Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bio-K Plus International Inc. (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111005-SCN-BIO-IBS-RA
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2015-04

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic capsules (Active Comparator): L. acidophilus CL1285® + L. casei LBC80R® + L. rhamnosus CLR2®. Dosage of 2 capsules per day , corresponding to 100 billions bacterias for a period of 12 weeks.
  Interventions: Dietary Supplement: L. acidophilus CL1285® + L. casei LBC80R® + L. rhamnosus CLR2®
- Placebo capsules (Placebo Comparator): The placebo capsules are identical in shape, taste, and smell yet are devoid of live bacteria. Dosage of 2 capsules per day , corresponding to 100 billions bacterias for a period of 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L. acidophilus CL1285® + L. casei LBC80R® + L. rhamnosus CLR2® — Each capsule contains 50 billion cfu live of Lactobacillus acidophilus CL1285® + L. casei LBC80R® + L. rhamnosus CLR2® bacterias. The randomized subjects will consume 2 capsules per day at breakfast.
  Other Names: Bio-K+
  Arms: Probiotic capsules
Other: Placebo — The placebo capsules are identical in shape, taste, and smell yet are devoid of live bacteria.
  Arms: Placebo capsules

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Bio-K+ on symptoms of IBS.

DETAILED DESCRIPTION:
Given the promising clinical results of previous trials of probiotics for IBS symptoms, the objective of this clinical trial is to evaluate the safety and effectiveness of a proprietary probiotic product, Lactobacillus acidophilus CL1285®, Lactobacillus casei LBC80R® and Lactobacillus rhamnosus CLR2® on symptoms of IBS in otherwise healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Subject meets Rome III criteria for IBS (regardless of IBS subtype) as follows:

   * Recurrent abdominal pain or discomfort at least 3 days/month in the last 3 months associated with 2 or more of the following:

     * Improvement with defecation
     * Onset associated with a change in frequency of stool
     * Onset associated with a change in form (appearance) of stool
   * Symptom onset must be at least 6 months prior to diagnosis
3. Agree to use contraception throughout study period, unless postmenopausal or surgically sterile (females only)
4. Able to understand the nature and purpose of the study including potential risks and side effects
5. Willing to consent to study participation and to comply with study requirements

   * Abdominal pain or discomfort at least 2 days during run-in period associated with 2 or more of the following:

     * Improvement with defecation
     * Onset associated with a change in frequency of stool
     * Onset associated with a change in form (appearance) of stool
   * Completion of all study-related questionnaires

Exclusion Criteria:

1. Diagnosed gastrointestinal disease, e.g. Crohn's disease, ulcer, cancer
2. Prior abdominal surgery that, in the investigator's opinion, may confound study outcomes
3. Any systemic disease that may confound IBS symptoms or compromise subject safety
4. Life expectancy < 6 months
5. Pregnant female or breastfeeding
6. Lactose intolerance
7. Immunodeficient subjects
8. Uncontrolled psychiatric disorder
9. Current treatment with nasogastric tube, ostomy, or parenteral nutrition
10. Eating disorder
11. Recent (< 2 weeks) antibiotic administration
12. History of alcohol, drug, or medication abuse
13. Daily consumption of probiotics, fermented milk, and/or yogurt
14. Known allergies to any substance in the study product
15. Participation in another study with any investigational product within 3 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
IBS Adequate Relief (IBS-AR) | 12 weeks
  The IBS-AR is a single-question dichotomous (yes/no) tool that asks subjects if they have experienced adequate relief of IBS symptoms over the past week.

SECONDARY OUTCOMES:
IBS Global Assessment of Improvement Scale | 12 weeks
  The IBS-GAI tool asks a single question regarding how recent IBS symptoms have changed since the start of the study. Subjects answer the question on a 1-7 Likert scale with 1 corresponding to "Substantially Worse" and 7 corresponding to "Substantially Improved".
IBS Symptom Severity Scale | 12 Weeks
  The IBS-SSS is a 5-question survey that asks the severity of abdominal pain, frequency of abdominal pain, severity of abdominal distention, dissatisfaction with bowel habits, and interference with quality of life over the past 10 days. Subjects respond to each question on a 100-point visual analogue scale
IBS Quality of Life | 12 Weeks
  The IBS-QOL is a 34-item questionnaire that assesses the degree to which IBS interfered with quality of life for a subject over the past 30 days. Each item is rated on a 1 to 5 Likert scale, with higher values indicating a lower quality of life.
Abdominal Pain | 12 Weeks
  Abdominal pain severity will be measured on a 0-10 Likert scale.
Stool Consistency | 12 Weeks
  Stool consistency will be rated with the Bristol Stool Chart.
Stool frequency | 12 Weeks
  Throughout the study, subjects will record the number of defecations per day in a diary.
Concomitant medication use | 12 Weeks
  Throughout the study, subjects will record use of any concomitant medication and, if required, the need for rescue medication use each day in a diary.
Adverse Events | 12 Weeks
  Adverse events will be assessed throughout this clinical study. The main safety endpoint will be the proportion of subjects in each group that report one of more AEs at any time during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Perelman, MS,RD,CDE, Principal Investigator — SPRIM ALS; Syam P. Gaddam, MD, Principal Investigator — Digestive and Liver Disease Specialists A medical Group Inc.; Razming Krumian, DO, Principal Investigator — Westlake Medical Research
Locations (3):
- United States (3):
  - Digestive and Liver Disease Specialists A Medical Group. Inc, Garden Grove, California
  - Sprim ALS, San Francisco, California
  - Westlake Medical Research, Westlake Village, California